CLINICAL TRIAL: NCT03811431
Title: Real Time Contrast-enhanced Compared to Conventional Ultrasound Guided Biopsy in the Diagnosis of Hepatic Tumors on a Background of Advanced Chronic Liver Disease. A Prospective Clinical Study.
Brief Title: Contrast Enhanced Ultrasound Guidance Biopsy for the Diagnosis of Liver Tumors
Acronym: ConCLUDe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Tudor Mocan, MD Associate Specialist, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: BIOPTICON
Record Dates: First submitted 2019-01-16; First posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Liver Diseases
Keywords: contrast enhanced ultrasound guided liver biopsy; ultrasound guided liver biopsy; focal liver lesions; hepatocellular carcinoma; advanced chronic liver disease
MeSH Terms: conditions — Liver Diseases; Carcinoma, Hepatocellular | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: A prospective parallel group clinical trial
Who Masked: Participant, Investigator
Masking Description: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CEUS guidance (Experimental): SonoVue 2, 4 ml
  Interventions: Procedure: Contrast enhanced ultrasound guided liver biopsy
- Conventional US guidance (Experimental): No drugs
  Interventions: Procedure: Contrast enhanced ultrasound guided liver biopsy

INTERVENTIONS:
Procedure: Contrast enhanced ultrasound guided liver biopsy — Conventional liver biopsy
  Other Names: Ultrasound

SUMMARY:
The main purpose of this study is to compare contrast-enhanced ultrasound guided liver biopsy (CEUS-LB) with conventional ultrasound guided liver biopsy (US-LB) in the diagnosis of liver tumors developed on a background of advanced chronic liver diseases. All patients referred to our department with a CT/MRI diagnosis of hepatic neoplasia will be randomly assigned to either CEUS-LB or US-LB. All LB will be performed by the same investigator. For the randomisation the flip coin technique will be used. One investigator without access to previous C/MRI/US report will do the randomization

DETAILED DESCRIPTION:
A prospective parallel group clinical trial will be performed. The study protocol was implemented in our Institute starting January 2011 ending January 1 2020. During this period, all patients with a suspicion of primary liver neoplasia either on CT or MRI will be evaluated in different departments from our Institute for possible inclusion. Patients with a typical aspect of benign FLLs will not be included in the study. Patients fulfilling the following criteria: presence of cirrhosis or other chronic liver disease (according to a liver stiffness evaluated by transient elastography higher than 10 kilopascals), Child-Pugh score no higher than B7 and absence of perihepatic ascites, platelet count > 50.000 per mm3 or an international normalized ratio < 1.6; will be further on sent to the department of interventional ultrasound. ). All patients referred to interventional department will underwent a B-mode ultrasound (1 investigator) testing the feasibility of performing liver biopsy. At this time point the conspicuity of the tumors will be recorded into either poorly or not poorly visible. Included patients will be randomly divided by another investigator (T.M.) without access to the previous US, CT or MRI report into two groups: a group that will underwent US guided liver biopsy (USLB) and another one who will underwent CEUS guided liver biopsy (CEUSLB). The randomization will be made based of flip coin technique. The side of the coin (heads-USLB, tails CEUSLB) determined the assignment of each subject. All biopsies will be performed by the same investigator (Z.S.) with an experience of more than 8 years in ultrasound interventions. Patients assigned to USLB or CEUSLB will be blinded. The investigators assessing the outcomes will not be informed about the LB technique used in each patient. The reasons for performing biopsy will be either inconclusive CT/MRI findings , or patients with a typical pattern of HCC on CT/MRI in whom a histological diagnosis is necessary in order to start systemic therapy (sorafenib). Different from other major society's guidelines, in our country a histological diagnosis of HCC is mandatory in patients referred for sorafenib treatment. Patients with small FLLs (BCLC 0 or A) and typical aspect of HCC on CT/MRI will be sent directly to surgery or radiofrequency ablation according to EASL guidelines.

ELIGIBILITY:
Inclusion Criteria:

* presence of cirrhosis or other chronic liver disease (according to a liver stiffness evaluated by transient elastography higher than 10 kilopascals)
* Child-Pugh score no higher than B7 and absence of perihepatic ascites
* platelet count > 50.000 per mm3
* international normalized ratio < 1.6

Exclusion Criteria:

* tumors located tin sonography blind areas
* refuse to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients in whom contrast enhanced ultrasound guided liver biopsy leads to the final diagnosis as compared to conventional ultrasound guided liver biopsy. The final diagnosis will be assessed based on histological examination. | From randomisation until the first documented histological diagnosis. In cases with a negative diagnosis based on histology imaging follow-up using CT or MRI will be carried on for a period of at least 12 months.
  In patients in whom a final histological diagnosis can not be achieved with the use of contrast enhanced or ultrasound guidance a second liver biopsy will be considered if appropriate in the next 3-4 weeks. In cases where a second liver biopsy will be judged not to be necessary a follow-up using imaging techniques will be performed until a final diagnosis is reached.

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Institute of Gastroenterology and Hepatology "Octavian Fodor", Cluj-Napoca, Please Enter the State Or Province, Romania

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data available within 12 months of study completion
Access Criteria: Data access request will be reviewed by an external Independent review panel.